CLINICAL TRIAL: NCT03293797
Title: Improving Access to Quality Mental Healthcare Through Innovations in Psychotherapy: A Pilot Study of a Novel, Ultra-Brief Intervention to Reduce Depressive and Anxious Symptoms
Brief Title: Ultra-Brief Intervention to Reduce Depressive and Anxious Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 387-2015
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Anxiety; Depression; Mood
Keywords: Mindfulness-based Therapy; Wellbeing; Treatment
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abbreviated Mindfulness-based Therapy (Experimental): 5 week, abbreviated group MBT treatment for depression and anxiety
  Interventions: Behavioral: Abbreviated-Mindfulness-based Therapy

INTERVENTIONS:
Behavioral: Abbreviated-Mindfulness-based Therapy — A-MBT will be delivered in group format, 120 minutes per week, for 5 consecutive weeks with 10-20 participants per group.
  Other Names: A-MBT

SUMMARY:
Symptoms of depression and anxiety are extremely prevalent in the population. Unfortunately, patients often face barriers to accessing mental health care, particularly psychotherapeutic interventions, including long wait-times and demanding therapeutic protocols. For instance, Mindfulness-Based Therapy (MBT) has demonstrated effectiveness at decreasing symptoms of depression and anxiety, and improving wellbeing; however, 'traditional' MBT can demand over 30 hours of clinical time, and 50-60 hours of homework, all of which can be barriers to care. A pilot, uncontrolled study conducted at Sunnybrook illustrated the potential feasibility / efficaciousness of a novel abbreviated MBT in improving hospital staff wellbeing. The goal of this controlled study is to further test feasibility and acceptability of this intervention to reduce depressive / anxious symptoms, reduce stress and improve wellbeing in outpatient mood/anxiety patients. If efficacious, this Abbreviated MBT could reduce barriers to accessing mental health care.

DETAILED DESCRIPTION:
BACKGROUND: ABBREVIATED-MINDFULNESS BASED THERAPY (A-MBT)

By the age of 40, 1 in 2 Canadians have been or are presently experiencing mental health issues. In particular, anxiety and mood disorders are the most prevalent lifetime mental health illnesses, affecting 11.6% of the population. Mindfulness based treatments (MBTs) have strong evidence for improving patient wellness through reduction of anxiety and mood symptoms in clinical populations. Although efficacious, 'traditional' MBTs are very demanding in terms of time and homework a relevant factor when considering the recent calls for waittime reductions in psychotherapeutic mental health services. These programs take 30+ hours (including 2-3 hr. weekly sessions across 8 weeks, plus a 1-day retreat) and expect 45-60 min./day of meditation homework. The goal of this project is to test the effectiveness of an abbreviated MBI in reducing anxiety and/or mood disturbances and improving patient well-being.

MBTs use a non-stigmatizing approach, combining secularized eastern meditative practices with western psychological advances to improve stress-management and self-care. Participants learn to generate less distress, engage more positively and fully in their lives and experiences, and respond more adaptively to challenges instead of reacting in automatic and unhelpful ways. Participants in MBI often describe the intervention as transformative. Professional experience and new insights into MBTs suggest that these 'tradition' treatment programs can be further abbreviated to develop a effective and accessible clinical intervention. This abbreviated MBT has been developed, which if effective will curtail wait-times and increase patient treatment annually.

RATIONAL & HYPOTHESIS/RESEARCH QUESTION Rational

Patients face barriers to accessing psychotherapy, including long wait-times and/or protocols that are too demanding for many patients. Traditional Mindfulness-Based Therapies (MBTs) are highly studied and well-recognized treatment options to reduce anxiety and mood symptoms - demonstrating repeated efficacy in clinical populations. However, the high demands of clinical time and homework are a barrier to many patients. Further, longer clinical interventions mean fewer patients being treated per hour of clinician's time, and therefore longer wait-times. Clinical experience and new insights into MBTs suggest that these 'tradition' treatment programs can be further abbreviated to develop an effective and more accessible therapy. If this Abbreviated MBT is demonstrated to be clinically effective, it can reduce barriers to mental health care by reaching more patients in a more timely fashion.

The specific objective of this study will be to evaluate a novel and potentially highly effective strategy to reduce depressive / anxious symptoms and stress, while improve quality of life and mental wellbeing among mood and anxiety outpatients referred to the Mindfulness-Based Therapy Clinic at Sunnybrook Health Sciences Centre.

Hypothesis/Research Question The study hypothesis is that an abbreviated MBT for mood / anxiety outpatient populations will show improvement in self-reported measures of clinical primary (Depression, Anxiety) and secondary (well-being, stress, self-compassion) outcomes and will be feasible for the population. Feasibility will be determined by patient program adherence (70% of participants attend ≥75% of sessions) and effect size (moderate magnitude of change in PHQ-9 / GAD-7), Cohen's d = ≥0.5). The effect size will provide a measure of how practically and clinically significant the treatment effect is, by measuring change in baseline, pre-treatment, post-treatment, 1/3/6 month and 1 year follow-up mean scores for the outcome measures.

Study Significance

The current pilot study will explore the effects of an Abbreviated-MBT on symptoms of depression and anxiety in an outpatient clinical sample; if effective: a) this would be the first known pilot study to consider and demonstrate efficacy of an Abbreviated-MBT in a clinical outpatient population; b) this treatment could increase the volume of patients treated by up to 3x, reduce wait-times by 2-3 fold, and reach a broader group of patients, including those for whom the investment of time of traditional MBT is too prohibitive

ELIGIBILITY:
Inclusion Criteria:

* Consenting mood and anxiety outpatients referred to Dr. Selchen in the Sunnybrook Mindfulness-Based Therapy Clinic
* Due to the nature of the assessment procedures, which include English-language self- report questionnaires and scales, ability to communicate in written and spoken English is an inclusion criterion

Exclusion Criteria:

* Patients who have active or recent (within 3 months) substance abuse/dependence, a history of dementia, untreated posttraumatic stress symptoms, active psychotic or manic symptoms, recent suicide attempt/active suicidality, or current self-injurious behaviour
* Previously completed a course (≥ 8 weeks) of a Mindfulness-Based Therapy within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptoms at 5 Week | Baseline (Week 0), Pre- (Week 1) and Post-Treatment Assessment (Week 5)
  Scale used to measure Depressive Symptoms: Patient Health Questionnaire 9-item (PHQ-9)
Change from Baseline Anxiety Symptoms at 5 Week | Baseline (Week 0), Pre- (Week 1) and Post-Treatment Assessment (Week 5)
  Scale used to measure Anxiety Symptoms: Generalized Anxiety Disorder 7-item (GAD-7)

SECONDARY OUTCOMES:
Change from Baseline Mental Wellbeing at 5 Week | Baseline (Week 0), Pre- (Week 1) and Post-Treatment Assessment (Week 5)
  Scale used to measure Mental Wellbeing: Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS)
Change from Baseline Self-Compassion at 5 Week | Baseline (Week 0), Pre- (Week 1) and Post-Treatment Assessment (Week 5)]
  Scale used to measure Self-Compassion: Self-Compassion Scale Short-Form (SCS-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Selchen, MD MSt FRCPC, Principal Investigator — Sunnybrook Healthy Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided